CLINICAL TRIAL: NCT04000971
Title: C3FIT (Coordinated, Collaborative, Comprehensive, Family-based, Integrated, Technology-enabled Care): A Randomized Trial for Stroke
Brief Title: Coordinated, Collaborative, Comprehensive, Family-based, Integrated, Technology-enabled Stroke Care
Acronym: C3FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kenneth Gaines, Professor, Neurology; Medical Director, Vanderbilt Teleneurology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: C3FIT
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Stroke, Ischemic; Stroke, Acute; Stroke Sequelae; Engagement, Patient; Stroke Hemorrhagic
Keywords: Technology-enabled; Engagement, caregiver; Team-based; Integrated Care
MeSH Terms: conditions — Stroke; Ischemic Stroke; Patient Participation; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized trial of approximately 22 clinical sites in the United States; randomization is by clinical site.
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes will be assessed by telephone at 3, 6, and 12 months by the University of Alabama at Birmingham (UAB)'s Survey Research Unit (SRU). Research staff at the SRU will be masked to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Stroke Practice Unit (ISPU) (Active Comparator): ISPU personnel will continue with care provided under the Joint Commission-certified CSC/PSC design, including a 30-day clinic visit post-discharge. This will be supplemented by a more integrated model designed to increase coordination through team-based initiatives across the continuum of care for stroke - from acute and in-hospital care through 12 months post-discharge. Care teams will follow patients in their home or rehabilitation/skilled nursing facility monthly for 12 visits to assess recovery, manage risk factors, increase understanding, and build positive behavior change for patients and caregivers. Primary outcomes will be assessed by phone at 3, 6, and 12 months; secondary outcomes will be assessed at 3, 6, and 12 months.
  Interventions: Other: Integrated Stroke Practice Unit
- Comprehensive or Primary Stroke Center (CSC/PSC) (Active Comparator): CSC/PSC personnel will continue with care provided under the Joint Commission-certified CSC/PSC design, including a 30-day clinic visit post-discharge, follow-up clinic visits as recommended by their outpatient provider, and other clinic visits initiated by the patient when issues arise. Primary outcomes will be assessed by phone at 3, 6, and 12 months; secondary outcomes will be assessed at 3, 6, and 12 months.
  Interventions: Other: Comprehensive or Primary Stroke Center

INTERVENTIONS:
Other: Integrated Stroke Practice Unit — Care teams will follow patients in their home or rehabilitation/skilled nursing facility monthly for 12 visits to assess recovery, manage risk factors, and increase understanding and build positive behavior change for patients and caregivers. Primary and secondary outcomes will be assessed at 3, 6, and 12 months.
  Other Names: ISPU
  Arms: Integrated Stroke Practice Unit (ISPU)
Other: Comprehensive or Primary Stroke Center — Primary and secondary outcomes will be assessed at 3, 6, and 12 months.
  Other Names: CSC/PSC
  Arms: Comprehensive or Primary Stroke Center (CSC/PSC)

SUMMARY:
Stroke is the 5th leading cause of death and the leading cause of adult disability in the United States (US). Stroke is a complex disease with multiple interacting risk factors (including genetic, high blood pressure and cholesterol, and lifestyle factors like smoking, diet, and exercise) that lead to initial and recurrent stroke. Up to 90% of stroke survivors have some functional deficit that impacts both physical and mental health.

Scientific evidence that identifies the best stroke care delivery design is lacking. We completed a three-year, Centers for Medicare & Medicaid Services (CMS) Health Care Innovation Award that tested a new stroke care design called an Integrated Practice Unit (IPU). This IPU was developed through stakeholder input from patients, caregivers, nurses, stroke specialists, rehabilitation specialists, patient advocacy groups, payers, and technology companies. This IPU design was associated with decreased hospital length of stay, readmissions, and stroke recurrence, as well as lower cost.

Based on the CMS study, a larger, pragmatic trial was developed that is called C3FIT (Coordinated, Collaborative, Comprehensive, Family-based, Integrated, and Technology-enabled Stroke Care). C3FIT will randomly assign approximately 22 US hospital sites to continue Joint Commission-certified Comprehensive/Primary (CSC/PSC) design or to the novel Integrated Stroke Practice Unit (ISPU) design for stroke care. C3FIT's ISPU uses team-based, enhanced collaboration (called Stroke Central) and follows patients from presentation at the Emergency Department (ED) through 12-months post-discharge (called Stroke Mobile). Stroke Mobile includes a nurse and lay health educator team who visit patients and caregivers at home or at a rehabilitation or skilled nursing facility to assess function and quality of life using telehealth technology to facilitate access to multiple providers. Results from C3FIT will provide high quality scientific evidence to determine the best stroke care design that ensures positive health for patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+.
* Clinical diagnosis of acute stroke with brain imaging compatible with intracerebral hemorrhage or ischemic stroke (including normal brain scan); see ICD 10 codes.
* English or Spanish speaking subjects.
* Patient admitted within 7 days of their index stroke event.
* Patient is discharged alive and not to hospice care.
* Patient living at discharge within the geography of recruitment for that C3FIT site.
* Pre-morbid mRS Rankin score of 0-1.
* Patient and/or surrogate give consent to participate after an informed consent process.
* Patients who go to rehabilitation inpatient therapy or other care facilities are eligible, as long as they reside in the geographic are of recruitment and do not go to hospice care.

Exclusion Criteria:

* Clinical transient ischemic attack (TIA)38-41 is excluded even if there is a computerized tomography (CT) or magnetic resonance imaging (MRI) lesion corresponding to the clinical syndrome at presentation.
* Already enrolled or planned enrollment in another clinical trial for which participation in C3FIT would be compromised with regard to follow-up assessment of outcomes or continuation in C3FIT.
* Patients with a planned admission to hospice care prior to consent.
* Patients not anticipated to survive for 1-year due to neurological or other medical status (i.e., advanced cancer, hospice care, heart disease, etc.).
* Patients who in the opinion of the site investigator cannot be involved in follow up care.
* Inability or unwillingness of subject or legal guardian/representative to understand and cooperate with study procedures or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale (SIS 3.0) | 12 months post-stroke
  59-item questionnaire to assess aspects of patient quality of life following stroke; includes 8 dimensions assessed on a 5-point Likert scale that are summed by domain. Scores range from 0-100, with higher scores indicating less difficulty.
Modified Rankin Scale | 12 months post-stroke
  7-item scale to assess the degree of disability/dependence in the daily activities of stroke patients; scores range from 0-5, with higher score indicating higher disability (a score of 6 indicates that the patient expired).

SECONDARY OUTCOMES:
Stroke Impact Scale 3.0 | 3 and 6 months post-stroke
  59-item questionnaire to assess aspects of patient quality of life following stroke; includes 8 dimensions assessed on a 5-point Likert scale that are summed by domain. Scores range from 0-100, with higher scores indicating less difficulty.
Modified Rankin Scale | 3 and 6 months post-stroke
  7-item scale to assess the degree of disability/dependence in the daily activities of stroke patients; scores range from 0-5, with higher score indicating higher disability (a score of 6 indicates that the patient expired).
Stroke Risk Factors - Blood Pressure Control (BP) | 3, 6, and 12 months post-stroke
  To assess BP control through measurement of a seated patient using a blood pressure cuff; controlled BP is 120-130/80 or below for ischemic stroke patients and 140/80 or below for hemorrhagic stroke patients.
Stroke Risk Factors - Cholesterol (LDL) | 3, 6, and 12 months post-stroke
  To assess LDL/lipids control through a LDL or lipids blood draw (standard of care) for patients with elevated cholesterol at baseline (prior to hospital discharge); controlled LDL is less than/equal to 70 for stroke patients.
Stroke Risk Factors - Blood Sugar (HgBA1c) | 3, 6, and 12 months post-stroke
  To assess blood sugar control through a HgBA1c blood draw (standard of care) for patients with elevated blood sugar at baseline (prior to hospital discharge); controlled HgBA1c is less than/equal to 7% for stroke patients.
Stroke Risk Factors - Body Mass Index (BMI) | 3, 6, and 12 months post-stroke
  To assess weight status by measuring patients' weight and height and applying a formula; patients with normal weight have BMI=18.5-24.9 (BMI less than 18.5 is underweight, and BMI 25.0 or above is overweight (BMI=25.0-29.9) or obese (BMI=30.0 or above).
Stroke Risk Factors - Smoking Status/Cessation | 3, 6, and 12 months post-stroke
  To assess smoking status and cessation efforts through self-reported, yes or no questions.
Stroke Risk Factors - Diet | 3, 6, and 12 months post-stroke
  To assess awareness of the DASH or Mediterranean diet through self-reported, yes or no questions.
Stroke Risk Factors - Exercise | 3, 6, and 12 months post-stroke
  To assess adherence to exercise guidelines that physician or physical therapist advised through self-reported, yes or no questions.
Mortality | 3, 6, and 12 months post-stroke
  Mortality following stroke will be assessed with family member, through study personnel, and/or using public sources.
Recurrence | 3, 6, and 12 months post-stroke
  Recurrence of stroke will be assessed/confirmed with study personnel.
Rehospitalization | 3, 6, and 12 months post-stroke
  Rehospitalization following stroke will be assessed/confirmed with study personnel.
Time at Home | 3, 6, and 12 months post-stroke
  Time spent at home compared to institution will be assessed/confirmed with study personnel.
Depression: Patient Health Questionnaire (PHQ-9) | 3, 6, and 12 months post-stroke
  9-item questionnaire to assess presence and/or severity of patient depression (includes an additional question to assess difficulty that doesn't impact scoring); scores range from 0-27, with 0=No depression, 1-4=Minimal depression, 5-9=Mild depression, 10-14=Moderate depression, 15-19=Moderately severe depression; and 20-27=Severe depression.
Modified Caregiver Strain Index (mCSI) | 3, 6, and 12 months post-stroke
  13-item questionnaire to assess the level of strain in caregivers; scores range from 0-100, with higher score indicating increased caregiver strain.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Gaines, MD, Principal Investigator — Vanderbilt University Medical Center; Barry Jackson, Principal Investigator; George Howard, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Emory University/Grady Health, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Intermountain, Las Vegas, Nevada
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Ohio Health Riverside Methodist Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Penn State, State College, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Johnson City Medical Center at Ballad Health, Johnson City, Tennessee
  - Covenant Health Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Doctors Hospital Renaissance, Edinburg, Texas
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Commiskey P, Long DL, Howard VJ, Braunlin J, Howard G, Cochran D, Jackson B, Bell D, Hill D, Callahan AE, Gaines K. Design and methods of a cluster-randomized pragmatic trial of post-discharge stroke care. Contemp Clin Trials. 2025 Jun;153:107890. doi: 10.1016/j.cct.2025.107890. Epub 2025 Apr 4. PMID 40189199